CLINICAL TRIAL: NCT05607329
Title: Secondary Cytoreduction Followed by Chemotherapy Versus Chemotherapy Alone in Relapsed Ovarian Cancer After PARPi Maintenance Treatment: a Multicenter, Open-label, Randomized, Phase 3 Trial
Brief Title: Secondary Cytoreduction Followed by Chemotherapy Versus Chemotherapy Alone in Relapsed Ovarian Cancer After PARPi Maintenance Treatment: a Multicentre, Open-label, Randomised, Phase 3 Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Women's Hospital School Of Medicine Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCAP-3
Record Dates: First submitted 2022-11-02; First posted 2022-11-07 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-01

CONDITIONS: Relapsed Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Secondary cytoreduction followed by chemotherapy (Experimental)
  Interventions: Procedure: Secondary cytoreduction; Drug: Chemotherapy
- chemotherapy alone (Active Comparator)
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Procedure: Secondary cytoreduction — Open surgery is conducted by senior clinicians in gynecological oncology. Operation time，location and number of relapsed lesions, location and number of excised lesions, Whether achieved R0 or not, and other information are recorded.
  Arms: Secondary cytoreduction followed by chemotherapy
Drug: Chemotherapy — chemotherapy

SUMMARY:
This study aims to carry out a multi-center, randomized controlled study on patients with recurrent ovarian cancer after PARPi maintenance, to explore the clinicopathological and molecular characteristics of patients with recurrent ovarian cancer after PARPi maintenance, and to clarify whether patients with recurrent ovarian cancer after PARPi maintenance for more than 6 months are sensitive to platinum drugs, and the value of secondary tumor cell reduction in such treatment, In order to provide evidence-based medicine basis for the standardized treatment mode of recurrent ovarian cancer after PARPi maintenance treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with diagnosis of first-line or second-line recurrent epithelial ovarian carcinoma, peritoneal carcinoma, or fallopian tube carcinoma, who has previously received at least 4 cycles of platinum-based chemotherapy in initial treatment;
2. Relapse occurred after 6 month since platinum-based chemotherapy;
3. PARPi maintenance therapy for more than 6 months before relapse;
4. R0 ideal debulking in initial surgery;
5. PET-CT indicate the recurrence lesion is isolated and not exceed 5 sites, and the ascites is less than 500ml;
6. ECOG/WHO Performance score of 0 to 1;
7. No hepatic failure, bilirubin ≤ 1,5 time the Normal limit, ASAT and ALAT ≤ 3 time the Upper Normal Limit
8. No Renal insufficiency (serum creatinine < 1,5 time the normal limit, creatinine clearance > 80 mL/min). calculated with MDRD method
9. Hematology function: PNN ≥ 1,5x10⁹/L, platelets ≥ 100x10⁹/L
10. No contraindication to general anaesthesia for heavy surgery
11. Patients having read, signed and dated Informed consent before any study procedure

Exclusion Criteria:

1. Platinum-refractory/uncontrolled epithelial ovarian cancer;
2. Non-epithelial ovarian tumor, mucinous, serous-mucinous (mainly mucinous), malignant Brenner tumor, low-grade serous carcinoma, borderline tumor;
3. Suffering from other malignant tumors that have not achieved complete remission in the past 2 years;
4. Received radiotherapy within 2 weeks before the start of the study intervention;
5. General conditions cannot tolerate secondary cytoreduction;
6. Severe hypersensitivity reactions (≥ grade 3) to paclitaxel or platinum and/or any of its excipients.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
progression free survival (PFS) | 18-24 months
  progression free survival

CONTACTS AND LOCATIONS:
Locations (1):
- Women's Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

REFERENCES:
- [Derived] Chen T, Xu J, Xia B, Wang H, Shen Y. Secondary cytoreduction surgery for recurrent epithelial ovarian cancer patients after PARPi maintenance: A multicenter, randomized, controlled clinical trial. Int J Gynecol Cancer. 2024 Feb 5;34(2):328-331. doi: 10.1136/ijgc-2023-004978. PMID 38159938